CLINICAL TRIAL: NCT03505905
Title: A Neurosteroid Intervention for Menopausal and Perimenopausal Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sherwood Brown, MD, PhD, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102017-068
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder; Menopause; Perimenopause
Keywords: Pregnenolone
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Pregnenolone

STUDY DESIGN:
Intervention Model Description: A double-blind, placebo-controlled, Sequential Parallel Comparison Design (SPCD) trial of pregnenolone. SPCD is a clinical trial design that may reduce the effect of placebo response on signal detection and maximize the ability to assess efficacy by dividing the trial into two phases, and then re-randomizing placebo non-responders.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pregnenlone (phase 1 and 2) (Experimental): Participants will receive pregnenolone at phase 1 (baseline-WK 7) and 2 (WK 8-16). The titration schedule is as follows: at baseline a 50 mg (BID, 7 days). WK 1=150 mg (BID, 7 days); WK 2=250 mg (BID, 14 days) and WK 4=250 mg (BID, 14 days) (BID, 14 days). At phase 2 (WK 8) to maintain the double blind of rerandomization, treatment in all conditions recommence at a dosage frequency similar to phase 1. At WK 8=250 mg (BID, 7 days); at WK 9=250 mg (BID, 7 days); WK 10=250 mg (BID, 14 days) and WK 12=250 mg (BID, 14 days) . During the participants' final WK (16), they will be instructed to titrate down the treatment according to the following schedule: 150 mg (BID, 4 days) and 50 mg (BID, 4 days), discontinue.
  Interventions: Drug: Pregnenolone
- Placebo rerandom to placebo (Placebo Comparator): Participants will receive placebo at phase 1 (baseline-WK 7) & treatment response assessed (MADRS score reduced <50% at WK8). Nonresponders are rerandomized to receive either treatment at phase 2 (WK8-16).The titration schedule is as follows (dosage throughout is BID): at baseline placebo (7 days). At WK 1= placebo (7 days); at WK 2=placebo (14 days) and WK 4=placebo (14 days). Placebo nonresponders rerandomized to placebo: At WK 8=placebo (7 days);WK 9=placebo (7 days);WK 10=placebo (14 days) and WK 12=placebo (14 days). During the participants' final WK (16), they will be instructed to titrate down (done in order to maintain the double blind) the treatment according to the following schedule: placebo (4 days) and placebo (4 days), discontinue.
  Interventions: Drug: Placebo
- Placebo rerandom to pregnenolone (Experimental): Participants will receive placebo at phase 1 (baseline-WK 7) & treatment response assessed (MADRS score reduced <50% at WK8). Nonresponders are rerandomized to receive either treatment at phase 2 (WK8-16).The titration schedule is as follows (dosage throughout is BID): at baseline placebo (7 days). At WK 1=placebo (7 days); WK 2=placebo (14 days) & WK 4=placebo (14 days). Placebo nonresponders who are rerandomized to pregnenolone: At WK 8=250 mg (7 days);WK 9=250 mg (7 days);WK 10=250 mg (14 days) & WK 12=250 mg (14 days). During the participants' final WK (16), they will be instructed to titrate down the treatment according to the following schedule: 150 mg (4 days) and 50 mg (4 days), discontinue.
  Interventions: Drug: Pregnenolone; Drug: Placebo
- Placebo responsive cont placebo (Placebo Comparator): Participants will placebo throughout phase 1 (baseline- WK 7) & treatment response assessed (MADRS score reduced <50% at WK8). Responders continue to receive placebo at phase 2 (WK8-16).The titration schedule is as follows (dosage throughout is BID): at baseline placebo (7 days). At WK 1=placebo (7 days); WK 2=placebo (14 days) & WK 4=placebo (14 days). Placebo responders remain on placebo: At WK 8, placebo (7 days); WK 9=placebo (7 days); WK 10=placebo (14 days) & WK 12=placebo (14 days). During the participants' final WK (16), they will be instructed to titrate down (done in order to maintain the double blind) the treatment according to the following schedule: placebo= 4 days) and placebo=4 days, discontinue.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone — In a sequential parallel comparison design, in a double blind placebo controlled study, the efficacy of pregnenlone treatment relative to placebo in improving depression and anxiety symptoms, cognition, sleep, quality of life and vasomotor symptoms in preimenopausal and menopausal women with MDD.
  Arms: Placebo rerandom to pregnenolone; Pregnenlone (phase 1 and 2)
Drug: Placebo — In a sequential parallel comparison design, in a double blind placebo controlled study, the efficacy of pregnenlone treatment relative to placebo in improving depression and anxiety symptoms, cognition, sleep, quality of life and vasomotor symptoms in preimenopausal and menopausal women with MDD.
  Arms: Placebo rerandom to placebo; Placebo rerandom to pregnenolone; Placebo responsive cont placebo

SUMMARY:
HYPOTHESIS:

Pregnenolone administration will be associated with greater reduction in depressive symptom severity than placebo in women with current mMDD.

STUDY AIMS:

Primary Aim: Determine if pregnenolone is associated with greater reduction in depressive symptom severity than placebo in women with mMDD, as measured by MADRS.

Secondary Aims:

1. Determine if pregnenolone is associated with greater reduction in anxiety symptom severity than placebo in women with mMDD.
2. Determine if pregnenolone is associated with greater improvement in cognition than placebo in women with mMDD.
3. Determine if pregnenolone is associated with greater improvement in quality of life than placebo in women with mMDD.
4. Determine if pregnenolone is associated with greater improvement in vasomotor symptoms of menopause than placebo.

Mechanistic Aims:

1. Determine whether changes in neurosteroid levels with pregnenolone mediate clinical response.
2. Determine if baseline neurosteroid levels predict pregnenolone response.
3. Determine whether depressive symptoms, anxiety, sleep or vasomotor symptoms improve first. A crossed-lagged panel model will explore serial correlations between changes in outcome measures.

DETAILED DESCRIPTION:
Despite the introduction of new antidepressants, major depressive disorder (MDD) remains challenging to treat. Antidepressant effectiveness trials conducted suggest depression remission rates of only 15%-35%. Therefore, new antidepressants with mechanisms that move beyond norepinephrine and serotonin targets are greatly needed. Importantly, comorbid symptoms including anxiety, cognitive complaints and somatic symptoms often co-occur with depression and further impact functioning and quality of life.

The lifetime prevalence of MDD in women at > 20%, is approximately twice of that of men, with increased risk during the menopausal transition (perimenopause and early postmenopause). Hot flashes and other menopausal symptoms, such as cognitive symptoms and sleep dysregulation, affect up to 80% of women after perimenopause onset. Two large NIH-funded prospective epidemiological studies demonstrated an increased risk of onset of MDD during perimenopause (mMDD), with hormonal variability serving as a biomarker of risk of MDD. Short-term studies have demonstrated an augmentation benefit of estrogen and serotonin reuptake inhibitors can be used to target both mMDD and hot flashes. However, limited data from controlled trials suggest modest benefit for mMDD with standard antidepressants. Furthermore, due to safety concerns, many women prefer options other than estrogen replacement. Therefore, new and more effective treatments are needed for mMDD. Despite the fact that midlife women are the most frequent consumers of complementary and alternative therapies, trials of these approaches for mMDD are lacking. Pregnenolone is a naturally occurring neurosteroid made from cholesterol in the adrenal glands and brain, sold as an over-the-counter supplement, and the use of which at this time is common, unregulated and unstudied in women around the menopausal transition. Pregnenolone is a precursor of hormones known to fluctuate during the menopausal transition, and may decrease this hormonal variability known to increase the risk of MDD.

Preclinical research suggests that pregnenolone has antidepressant and neuroprotective effects, and improves cognition. Lower cerebrospinal fluid levels of pregnenolone are reported in people with bipolar disorder (BPD) or major depressive disorder (MDD) than controls. The investigators conducted two pilot studies of pregnenolone in depressed patients. The first study included patients with bipolar as well as unipolar depression (i.e. MDD). Pregnenolone (100 mg/d) was superior to placebo in improving depressive symptom severity. The second study found that 500 mg/d of pregnenolone was superior to placebo for bipolar depression. Baseline anxiety, fatigue, anhedonia and physical symptoms predicted a favorable depressive symptom response to pregnenolone compared to placebo. Improvement in cognition (e.g. declarative and working memory) was also observed in women given pregnenolone. Additionally, in women, changes in depressive symptoms showed strong inverse correlations with changes in pregnenolone (r=-0.83), and other neurosteroid levels. Furthermore, in both studies women responded better to pregnenolone relative to placebo for depression than men. Therefore, pregnenolone appears to have sex-specific antidepressant effects, or at least demonstrates a substantial sex difference in response. Women over age 40 showed a more robust response than younger women. Pregnenolone was very well tolerated in both studies. Based on these data, a larger, longer and more definitive trial of pregnenolone is now proposed. Unlike the prior pilot studies, this trial will be larger and focus on unipolar rather than bipolar depression, and will be limited to women with mMDD.

Given the widespread availability of pregnenolone, as well as promising preclinical and clinical data, and the extensive use of integrative treatments among midlife women, the investigators propose to examine its efficacy as an antidepressant in mMDD. Pregnenolone has the potential to provide women with an efficacious and appealing treatment option. To achieve this objective, a randomized, placebo-controlled trial of pregnenolone is proposed in 144 women with mMDD. A novel clinical trial design that enhances power to detect between-group differences and that allows for a longer observation period (16 weeks) will be used. Depressive symptoms, anxiety, quality of life, cognition and vasomotor symptoms (e.g. hot flashes) will be assessed. Blood levels of pregnenolone, and other neurosteroids (e.g. allopregnanolone, progesterone) will be obtained, and safety and tolerability data collected. A multiple PI team with extensive experience in mood disorders clinical trials, women's mental health and neurosteroids will conduct the study.

ELIGIBILITY:
Inclusion Criteria:

The participants must meet the following criteria:

* Women aged 40-67 years who are perimenopausal or early postmenopausal (within 5 years of the last menstrual period if not surgically postmenopausal), including:
* Women who have experienced changes in menstrual cycle frequency or duration, and/or physical symptoms indicative of menopausal transition, as determined by clinician
* Women who are using hormonal IUDs (i.e. brands Mirena and Skyla), with FSH level > 20 mIU/m (as menstrual periods are irregular with IUDs that utilize hormones, making irregular/absent periods difficult to assess as related to the menopausal transition).
* Women with significant menopause-related physical symptoms, indicated by any of the following criteria:
* Greene Climacteric Scale total scores > 20
* Greene Climacteric Scale sub-score for vasomotor symptoms >3
* 5 or more bothersome hot flashes per week (self-reported)
* Women meeting DSM-5 criteria for current major depressive disorder (assessed by the SCID)
* Baseline HRSD score of ≥ 18
* Subject agrees to abstain from disallowed medications for the duration of the trial

Exclusion Criteria:

The participants must not meet any of the following criteria:

* Vulnerable populations (e.g. pregnant/nursing, severe cognitive or intellectual impairment, incarcerated)
* Pregnancy (determined by urine pregnancy test), intending pregnancy or breast feeding
* Psychiatric disorder other than MDD that is acute and the primary focus of symptom burden or treatment.
* History of bipolar disorder or psychotic disorder
* Current substance use disorder
* Positive baseline urine drug screen of an illicit substance (in this study: opioids and cocaine,) with the exception of a medication used with a prescription (use of a detected substance that is used with a prescription, such as an opioid pain medication, is not necessarily exclusionary and will be based upon judgment of the PI, particularly in the cases of chronic opioid use). Participants who screen positive for marijuana will be offered a rescreen for eligibility at a later date.
* Current eating disorder
* Treatment resistant depression (failure of 2 adequate antidepressant trials or electroconvulsive therapy (ECT) during current episode; adequate antidepressant trials are defined as within the US FDA approved dosage for the medication and used for at least 6 weeks, with failure described by the patient as <50% improvement based on her subjective experience).
* High risk for suicidal acts including active suicidal ideation with plan and intent or > 2 suicide attempts in lifetime or any attempt in the past 6 months
* Use of selective estrogen-receptor modulators (SERMs), hormone replacement therapy, hormonal contraceptives (hormonal IUDs allowed), episodic sleep medications (chronic, regular, stable-dose benzodiazepines and hypnotics such as zolpidem, Sonata (Zaleplon), and Lunesta (Eszopiclone) OR sleep-seating antihistamines such as Unisom (Doxylamine succinate) or diphenhydramine allowed) within 2 weeks of the baseline visit and randomization. Antidepressants will be allowed for those participants who have been taking the antidepressant for 6 weeks with a stable dose for at least 4 weeks.
* Use of natural menopause and depression supplements, phytoestrogens, soy-based medications, steroids within 2 weeks of baseline visit and randomization.
* Use of any disallowed medications (specified in the Excluded Concomitant Medication section below).
* Women who have received a gonadal hormonal intervention within 1 month prior to study entry (stable thyroid medications are allowed).
* Not using a medically approved method of birth control, if sexually active and not 12 or more months since last menstrual period IUDs, condoms, abstinence are acceptable forms of contraception in this study; due to the possible interactions with the study medication, oral contraceptive pills will be prohibited.
* Uncontrolled hypertension (>160/95mmHg)
* Active coronary artery disease, atrial fibrillation, stroke, deep vein thrombosis, pulmonary embolism or blood clotting disorder
* Any severe, life threatening or unstable medical condition that, based on clinician-judgment, would make participation in the study unsafe or inappropriate
* Personal or first degree family history of known hormone sensitive tumors
* History of allergic reaction or side effects with prior pregnenolone use
* Clinically significant laboratory or physical examination findings
* Concurrent enrollment in another clinical trial

Exclusion of Concomitant Medications:

* Selective estrogen-receptor modulators (SERMs)
* Hormone replacement therapy
* Hormonal contraceptives, excluding Mirena IUD or other IUD with localized progesterone
* Natural menopause or antidepressant supplements
* Episodic sleep medications (chronic, regular, stable-dose benzodiazepines and hypnotics such as zolpidem, Sonata (Zaleplon), and Lunesta (Eszopiclone) OR sleep-sedating antihistamines such as Unisom (Doxylamine succinate) or diphenhydramine allowed)
* Sub-therapeutic dosages of antidepressants used for other indications will be permissible with the exclusion of SSRIs, SNRIs, and Wellbutrin.
* Phytoestrogens
* Soy-based medications or supplements

Ages: 40 Years to 67 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center; Marlene Freeman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Pregnenolone - Pregnenolone: Phase 1 - Pregnenolone. Phase 2 - Pregnenolone.
  Group 1 includes participants who received pregnenolone in Phase 1 and in Phase 2. Group 1 also includes participants who received pregnenolone in Phase 1 but did not complete Phase 1 and thus did not start Phase 2. These participants were grouped here because, per Sequential Parallel Comparison Design (SPCD), participants who are randomized to receive pregnenolone in Phase 1 continue to receive pregnenolone in Phase 2.
- Group 2: Placebo - Pregnenolone: Phase 1 - Placebo. Phase 2 - Pregnenolone.
  Group 2 includes participants who received placebo in Phase 1, were non-responders, and were then re-randomized to receive pregnenolone in Phase 2. Per Sequential Parallel Comparison Design (SPCD), participants will be randomized to receive placebo or pregnenolone in a 2:1 ratio in Phase 1. Then, placebo non-responders in Phase 1 will be re-randomized in Phase 2 to receive placebo or pregnenolone in a 1:1 ratio.
- Group 3: Placebo - Placebo: Phase 1 - Placebo. Phase 2 - Placebo.
  Group 3 includes participants who received placebo in Phase 1, were non-responders, and were then re-randomized to receive placebo in Phase 2. Per Sequential Parallel Comparison Design (SPCD), participants will be randomized to receive placebo or pregnenolone in a 2:1 ratio in Phase 1. Then, placebo non-responders in Phase 1 will be re-randomized in Phase 2 to receive placebo or pregnenolone in a 1:1 ratio.
- Group 4: Placebo - No Phase 2: Phase 1 - Placebo. Phase 2 - Drop Outs & Placebo Responders.
  Group 4 includes participants who received placebo and dropped out in Phase 1 and did not proceed to Phase 2. Group 4 also includes all placebo responders regardless of whether they proceeded to Phase 2 since all placebo responders continue receiving placebo in Phase 2.
Period: Phase 1
Arm/Group | Group 1: Pregnenolone - Pregnenolone | Group 2: Placebo - Pregnenolone | Group 3: Placebo - Placebo | Group 4: Placebo - No Phase 2
Started | 26 | 9 | 7 | 31
Completed | 16 | 9 | 7 | 17
Not Completed | 10 | 0 | 0 | 14
Period: Phase 2
Arm/Group | Group 1: Pregnenolone - Pregnenolone | Group 2: Placebo - Pregnenolone | Group 3: Placebo - Placebo | Group 4: Placebo - No Phase 2
Started | 16 | 9 | 7 | 17
Completed | 14 | 8 | 6 | 15
Not Completed | 2 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Pregnenolone - Pregnenolone | Group 2: Placebo - Pregnenolone | Group 3: Placebo - Placebo | Group 4: Placebo - No Phase 2 | Total
Number analyzed (Participants) | 26 | 9 | 7 | 31 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 8 | 7 | 31 | 71
  >=65 years | 1 | 1 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.27 (6.87) | 52.78 (5.47) | 51.29 (6.32) | 50.42 (5.10) | 51.09 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 9 | 7 | 31 | 73
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 10 | 1 | 2 | 6 | 19
  White | 15 | 6 | 4 | 18 | 43
  More than one race | 1 | 0 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 7 | 11
  Not Hispanic or Latino | 23 | 8 | 7 | 24 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The Montgomery-Asberg Depression Rating Scale (MADRS; primary outcome) is an observer-rated 10-item measure of depressive symptomatology designed for use in clinical trials. Each item is rated from 0-6 in order of increasing severity based upon the assessment of symptoms within the past 7 days. The range of total scores is 0-60, with higher score indicative of more severe depressive symptoms.
Time Frame: Phase 1 timeframe is Baseline to Week 8; Phase 2 timeframe is Week 8 to Week 16
Population: Due to the methods used in Sequential Parallel Comparison Design (SPCD), Phase 2 analysis only includes participants who were placebo non-responders in Phase 1. The total number of participants who received pregnenolone in Phase 1 was 26 and the total number of participants who received placebo in Phase 1 was 47. Those who received pregnenolone in Phase 1 continued to receive Pregnenolone in Phase 2. Placebo responders in Phase 1 continued to receive placebo in Phase 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pregnenolone: Participants randomized to receive pregnenolone in Phase 1 continued to receive pregnenolone in Phase 2. The titration schedule was as follows: 50mg BID for 7 days at Baseline, 150mg BID for 7 days at Week 1, 250mg BID for 14 days at Week 2, and 250mg BID for 28 days at Week 4. Participants continued 250mg BID throughout Phase 2. At Week 16, participants titrated down at 150mg BID for 4 days and then 50mg BID for 4 days before discontinuing.
- Placebo: Participants received placebo at the same frequency as those who received pregnenolone. Placebo responders in Phase 1 continued to received placebo in Phase 2. Placebo non-responders in Phase 1 were rerandomized to receive either placebo or pregnenolone in Phase 2.
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 47
units on a scale
  Phase 1 - Baseline | 26.2 (5.0) | 27.0 (4.5)
  Phase 1 - Week 8: number analyzed (Participants) | 17 | 33
  Phase 1 - Week 8 | 15.7 (7.2) | 15.2 (8.7)
  Phase 1 - Change in Score: number analyzed (Participants) | 17 | 33
  Phase 1 - Change in Score | -11.8 (8.3) | -11.9 (8.6)
  Phase 2 - Week 8: number analyzed (Participants) | 9 | 7
  Phase 2 - Week 8 | 22.4 (7.4) | 22.1 (5.6)
  Phase 2 - Week 16: number analyzed (Participants) | 8 | 6
  Phase 2 - Week 16 | 14.4 (8.9) | 19.3 (5.6)
  Phase 2 - Change in Score: number analyzed (Participants) | 8 | 6
  Phase 2 - Change in Score | -8.8 (13.1) | -3.5 (6.0)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; Phase 1 analysis includes all randomized participants (n=73). Per SPCD, Phase 2 analysis only includes participants who were randomized to Placebo in Phase 1, and were non-responders in Phase 1 (n=16); Test type: Superiority; p = 0.29, Linear mixed effects model — No adjustment for multiple comparisons, as there was only one primary outcome variable; Phase 1 and 2 data are analyzed separately, and then combined for the overall treatment effect; Mean Difference (Final Values) = -2.4587 — Combined Phase 1 and 2 effect, based on the differences of the least squares means

2. Secondary Outcome: Hamilton Anxiety Rating Scale (HRSA)
Description: The Hamilton Anxiety Rating Scale (HRSA) is a 14-item observer-rated scale that assesses the degree and pathology associated with anxiety such as anxious mood, tension, fear, and insomnia. Items are scored 0 (absent) through 4 (very severe) with the total score ranging from 0 to 56. Higher scores indicate a greater degree of anxiety symptoms.
Time Frame: Phase 1 timeframe is Baseline to Week 8; Phase 2 timeframe is Week 8 to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 47
units on a scale
  Phase 1 - Baseline | 19.4 (5.1) | 19.2 (5.5)
  Phase 1 - Week 8: number analyzed (Participants) | 17 | 32
  Phase 1 - Week 8 | 14.5 (5.6) | 12.9 (5.3)
  Phase 1 - Change in Score: number analyzed (Participants) | 17 | 32
  Phase 1 - Change in Score | -5.2 (6.9) | -5.5 (5.3)
  Phase 2 - Week 8: number analyzed (Participants) | 9 | 7
  Phase 2 - Week 8 | 15.0 (3.9) | 16.3 (6.2)
  Phase 2 - Week 16: number analyzed (Participants) | 8 | 6
  Phase 2 - Week 16 | 13.3 (6.4) | 18.0 (4.9)
  Phase 2 - Change in Score: number analyzed (Participants) | 8 | 6
  Phase 2 - Change in Score | -2.3 (4.5) | 0.8 (4.8)

3. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a 9-item self-report scale used to assess sleep quality and disturbances during the past week. Total scores range from 0 to 21 with higher scores indicating poorer sleep quality. Total scores are calculated by adding together the scores of the 7 components (e.g., duration of sleep, sleep disturbance, sleep latency) that comprise the PSQI.
Time Frame: Phase 1 timeframe is Baseline to Week 8; Phase 2 timeframe is Week 8 to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 47
units on a scale
  Phase 1 - Baseline: number analyzed (Participants) | 24 | 47
  Phase 1 - Baseline | 7.5 (5.7) | 8.1 (4.0)
  Phase 1 - Week 8: number analyzed (Participants) | 16 | 32
  Phase 1 - Week 8 | 5.8 (4.9) | 6.2 (4.4)
  Phase 1 - Change in Score: number analyzed (Participants) | 14 | 32
  Phase 1 - Change in Score | -2.9 (4.5) | -2.5 (3.9)
  Phase 2 - Week 8: number analyzed (Participants) | 9 | 7
  Phase 2 - Week 8 | 7.1 (4.6) | 7.1 (6.0)
  Phase 2 - Week 16: number analyzed (Participants) | 8 | 6
  Phase 2 - Week 16 | 3.4 (1.6) | 5.5 (4.7)
  Phase 2 - Change in Score: number analyzed (Participants) | 8 | 6
  Phase 2 - Change in Score | -4.1 (3.9) | -0.5 (2.9)

4. Secondary Outcome: Menopause Specific Quality of Life (MEN-QOL)
Description: The Menopause Specific Quality of Life (MEN-QOL) is a 29-item measure used to assess the presence and bother associated with 29-different menopausal symptoms. Items are scored 0 (not bothered at all) to 6 (extremely bothered) with total scores ranging from 0 to 174. Higher total scores indicate worse menopausal symptoms.
Time Frame: Phase 1 timeframe is Baseline to Week 8; Phase 2 timeframe is Week 8 to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 47
units on a scale
  Phase 1 - Baseline: number analyzed (Participants) | 23 | 46
  Phase 1 - Baseline | 128.5 (32.1) | 141.0 (33.2)
  Phase 1 - Week 8: number analyzed (Participants) | 16 | 32
  Phase 1 - Week 8 | 83.3 (32.8) | 95.3 (35.4)
  Phase 1 - Change in Score: number analyzed (Participants) | 14 | 32
  Phase 1 - Change in Score | -61.4 (36.5) | -50.3 (30.3)
  Phase 2 - Week 8: number analyzed (Participants) | 9 | 7
  Phase 2 - Week 8 | 93.8 (35.3) | 104.1 (44.9)
  Phase 2 - Week 16: number analyzed (Participants) | 8 | 6
  Phase 2 - Week 16 | 78.0 (34.2) | 105.8 (41.0)
  Phase 2 - Change in Score: number analyzed (Participants) | 8 | 6
  Phase 2 - Change in Score | -16.9 (25.0) | -8.0 (24.9)

5. Secondary Outcome: Greene Climacteric Scale (GCS)
Description: The Greene Climacteric Scale (GCS) is a 21-item menopause symptom checklist providing an objective measure of mood disturbance, hot flushes, night sweats, and vaginal dryness. Items are scored from 0 (not at all) to 3 (extremely) with total scores ranging from 0 to 63. Higher total scores indicate worse menopause symptoms. Total scores are calculated by adding together the scores of the 3 subscales (e.g., psychological, vasomotor, physical) that comprise the GCS.
Time Frame: Phase 1 timeframe is Baseline to Week 8; Phase 2 timeframe is Week 8 to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 47
units on a scale
  Phase 1 - Week 8: number analyzed (Participants) | 23 | 43
  Phase 1 - Week 8 | 27.5 (10.2) | 31.4 (9.6)
  Phase 1 - End of Phase: number analyzed (Participants) | 15 | 29
  Phase 1 - End of Phase | 14.5 (8.0) | 13.7 (8.3)
  Phase 1 - Change in Score: number analyzed (Participants) | 13 | 27
  Phase 1 - Change in Score | -16.8 (8.3) | -16.7 (7.8)
  Phase 2 - Week 8: number analyzed (Participants) | 9 | 6
  Phase 2 - Week 8 | 15.9 (7.5) | 20.8 (10.2)
  Phase 2 - Week 16: number analyzed (Participants) | 7 | 5
  Phase 2 - Week 16 | 12.9 (9.0) | 20.8 (7.7)
  Phase 2 - Change in Score: number analyzed (Participants) | 7 | 5
  Phase 2 - Change in Score | -2.9 (6.9) | -2.0 (5.6)

6. Secondary Outcome: Rey Auditory Verbal Learning Test (RAVLT)
Description: The Rey Auditory Verbal Learning Test (RAVLT) is an auditory assessment of verbal learning and memory, in which the participant is asked to recall a list of words first immediately following presentation (immediate recall) and later following a set period of time (delayed recall). Participant age, years of education, and sex are used to calculate t-scores. T-scores represent how an individual score compares to the mean / average score of that participant's demographic group. Higher t-scores indicate a greater recall of the list of words compared to the average score.
Time Frame: Phase 1 timeframe is Baseline to Week 8; Phase 2 timeframe is Week 8 to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 47
units on a scale
  Phase 1 - Baseline: number analyzed (Participants) | 24 | 45
  Phase 1 - Baseline | 50.0 (10.3) | 51.3 (9.0)
  Phase 1 - Week 8: number analyzed (Participants) | 16 | 30
  Phase 1 - Week 8 | 53.3 (12.1) | 54.5 (14.4)
  Phase 1 - Change in Score: number analyzed (Participants) | 15 | 30
  Phase 1 - Change in Score | 2.9 (10.2) | 1.8 (13.7)
  Phase 2 - Week 8: number analyzed (Participants) | 8 | 7
  Phase 2 - Week 8 | 49.8 (20.2) | 59.0 (12.3)
  Phase 2 - Week 16: number analyzed (Participants) | 6 | 6
  Phase 2 - Week 16 | 57.5 (5.9) | 61.0 (9.5)
  Phase 2 - Change in Score: number analyzed (Participants) | 6 | 6
  Phase 2 - Change in Score | 9.0 (20.5) | 1.7 (6.3)

7. Secondary Outcome: Trail Making Test (TMT)
Description: The Trail Making Test (TMT) is a diagnostic tool measuring executive functioning and information processing in which the participant is asked to link a set of randomly distributed numbered and lettered points. Participant age, years of education, and sex are used to calculate t-scores. T-scores represent how an individual score compares to the mean / average score of that participant's demographic group. Higher t-scores indicate a faster time in connecting the set of numbers and letters compared to the average score.
Time Frame: Phase 1 timeframe is Baseline to Week 8; Phase 2 timeframe is Week 8 to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 47
units on a scale
  Phase 1 - Baseline: number analyzed (Participants) | 21 | 39
  Phase 1 - Baseline | 46.6 (11.4) | 51.5 (10.3)
  Phase 1 - Week 8: number analyzed (Participants) | 14 | 26
  Phase 1 - Week 8 | 56.6 (15.6) | 54.1 (10.7)
  Phase 1 - Change in Score: number analyzed (Participants) | 13 | 25
  Phase 1 - Change in Score | 8.3 (8.5) | 1.1 (9.8)
  Phase 2 - Week 8: number analyzed (Participants) | 7 | 7
  Phase 2 - Week 8 | 50.1 (9.5) | 51.0 (8.2)
  Phase 2 - Week 16: number analyzed (Participants) | 5 | 6
  Phase 2 - Week 16 | 56.8 (12.7) | 55.3 (9.2)
  Phase 2 - Change in Score: number analyzed (Participants) | 5 | 6
  Phase 2 - Change in Score | 3.8 (12.6) | 5.2 (1.8)

ADVERSE EVENTS:
Time Frame: The period of observation for the collection of adverse events extends from the time the subject gave informed consent until the final visit at Week 16.
Groups:
- Phase 1: Placebo: This group contains all participants who were randomized to receive Placebo in Phase 1.
- Phase 1: Pregnenolone: This group contains all participants who were randomized to receive Pregnenolone in Phase 1.
- Phase 2: Placebo: This group contains all participants who were randomized to receive Placebo in Phase 2.
- Phase 2: Pregnenolone: This group contains all participants who were randomized to receive Pregnenolone in Phase 2.
Arm/Group | Phase 1: Placebo | Phase 1: Pregnenolone | Phase 2: Placebo | Phase 2: Pregnenolone
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/26 | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/26 | 1/24 | 0/25
Other Adverse Events (participants affected / at risk) | 20/47 | 17/26 | 5/24 | 5/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Placebo (N=47) | Phase 1: Pregnenolone (N=26) | Phase 2: Placebo (N=24) | Phase 2: Pregnenolone (N=25)
Implant Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Placebo (N=47) | Phase 1: Pregnenolone (N=26) | Phase 2: Placebo (N=24) | Phase 2: Pregnenolone (N=25)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (4) | 0 (0)
Difficulty Falling Asleep (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 7 (7) | 4 (4) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 9 (10) | 5 (5) | 4 (4) | 4 (5)
Premenstrual Syndrome (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Ringing in Ear (Ear and labyrinth disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Heart Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Increased Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Increased Flatulence (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Nightmares (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Hot Flashes (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Increased Urinary Frequency (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT03505905/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT03505905/ICF_001.pdf